CLINICAL TRIAL: NCT07382570
Title: Multicenter Prospective Cohort Study Protocol on the Natural Course of Congenital Hydronephrosis in Infants Aged 0-6 Months (3-Year Cycle)
Brief Title: Natural Course of Congenital Hydronephrosis in Infants Aged 0-6 Months
Status: Not yet recruiting | Type: Observational
Sponsor: The Children's Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Principal Investigator, Guangjie Chen, Chief Physician, The Children's Hospital of Zhejiang University School of Medicine
Other Study IDs: 2026-IRB-0038-P-01
Record Dates: First submitted 2025-12-10; First posted 2026-02-03 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Congenital Hydronephrosis; UTD Grading System; Natural Progression; Pediatric

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- UTDⅠ
  Interventions: Other: No Intervention: Observational Cohort
- UTD II
  Interventions: Other: No Intervention: Observational Cohort
- UTD III
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — No intervention

SUMMARY:
This project aims to systematically delineate the natural progression of congenital hydronephrosis diagnosed within the critical window of 0-6 months through a prospective, multicenter, observational cohort study. The focus will be on analyzing the resolution rates, progression rates, and influencing factors of hydronephrosis of varying severities based on the UTD grading system.

Congenital hydronephrosis is one of the most common congenital urinary system abnormalities in children, with a high prenatal detection rate. However, its postnatal natural course is highly heterogeneous, leading to significant controversy in clinical management regarding follow-up intensity and intervention timing. Currently, there is a lack of prospective, large-sample, multicenter natural history data in China. By establishing a standardized follow-up system and collecting high-quality clinical and imaging data, this study aims to provide high-level evidence-based medical support for developing individualized and precise clinical management strategies, thereby reducing unnecessary interventions and delayed treatment. Consequently, conducting this multicenter study holds significant clinical and scientific value.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic Criteria: Congenital hydronephrosis is diagnosed by abdominal ultrasound examination and meets the UTD grading system criteria (Grades I-III). This is defined as an anterior-posterior renal pelvis diameter (APD) ≥4 mm during the fetal period or ≥7 mm after birth, or accompanied by calyceal dilation, renal parenchymal changes, and other manifestations.
* Informed Consent: The legal guardian voluntarily agrees to participate in the study and provides written informed consent.
* Follow-up Feasibility: The guardian commits to cooperating with the complete 3-year follow-up period, including attending regular examinations at the research center, and maintains stable contact information.

Exclusion Criteria:

* Presence of other severe congenital malformations that may affect follow-up or prognosis assessment, such as congenital heart disease, biliary atresia, spina bifida, etc.
* Secondary hydronephrosis caused by acquired factors (e.g., urinary system tumors, stones, trauma) or well-defined genetic metabolic diseases.
* Having received interventional treatments prior to enrollment, such as surgical procedures related to hydronephrosis (e.g., pyeloplasty) or pharmacological interventions (e.g., long-term use of diuretics).
* Severe underlying diseases that preclude tolerance for long-term follow-up, such as severe infections, respiratory failure, or renal failure (e.g., glomerular filtration rate < 30 ml/min/1.73m²).
* Inability of the legal guardian to cooperate due to mental illness, cognitive impairment, or refusal to comply with follow-up schedules and data collection requirements.

Ages: 0 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants diagnosed with congenital hydronephrosis by abdominal ultrasound within 0-6 months after birth, meeting the UTD classification criteria (Grades I-III).
Sampling Method: Non-Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Hydronephrosis Resolution Rate | During the follow-up period (3 years)
  During the follow-up period (3 years), the child's hydronephrosis decreased from the UTD grade at enrollment to grade I or below, and this status persisted for ≥6 months.

SECONDARY OUTCOMES:
Rate of Hydronephrosis Progression (UTD Classification) | During the follow-up period (3 years)
  Percentage of participants with an increase of ≥1 grade in the UTD classification compared to the baseline.
Rate of Renal Parenchymal Thinning | During the follow-up period (3 years)
  Percentage of participants with a decrease of ≥2mm in renal parenchymal thickness from baseline measured by ultrasound.
Incidence of Urinary Tract Infections (UTI) | During the follow-up period (3 years)
  The number of symptomatic UTI episodes per participant, characterized by a positive urine culture
Change in Estimated Glomerular Filtration Rate (eGFR) | During the follow-up period (3 years)
  The mean change from baseline in eGFR levels to assess the trend of renal function over time.
Change in Weight-for-age Z-score | During the follow-up period (3 years)
  The Z-scores are calculated based on the WHO Child Growth Standards to assess the child's weight development status.
Change in Height-for-age Z-score | During the follow-up period (3 years)
  The Z-scores are calculated based on the WHO Child Growth Standards to assess the child's linear growth development status.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's hospital, Zhejiang Univeristy School of Medicine, Hangzhou, Zhejiang, China